CLINICAL TRIAL: NCT05217329
Title: Smart Phone as an Assistive Technology for Stroke Upper Limb Motor Function Training - Feasibility and Treatment Effects Analysis
Brief Title: Smart Phone for Stroke Upper Limb Motor Function Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KMUHIRB-E(I)-20190067
Record Dates: First submitted 2022-01-24; First posted 2022-02-01 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2018-12

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- smart phone intervention group (Experimental): smart phone intervention group stroke subjects completed smart phone App tasks with affected arm or bilateral arm movement
  Interventions: Other: smart phone App rehabilitation
- conventional group (Active Comparator): stroke subjects receive conventional rehabilitation home program
  Interventions: Other: conventional rehabilitation

INTERVENTIONS:
Other: smart phone App rehabilitation — stroke subjects use smart phone to complete therapeutic tasks 5 min/session total 8 sessions/day with affected arm or bilateral arm movement for 6 weeks
  Arms: smart phone intervention group
Other: conventional rehabilitation — stroke subjects receive conventional rehabilitation home program for 6 weeks(30min/day)
  Arms: conventional group

SUMMARY:
Stroke rehabilitation for stroke patients can enhance the upper and lower limb function, daily of daily activity improvement, and be beneficial to the family members' quality of life. Literature studies have supported the use of tele-rehabilitation to be as effective as stroke home rehabilitation. Stroke tele-rehabilitation model can use smartphones and apps to practice the mobile health model. Nevertheless, effects of tele-rehabilitation analysis for the proximal recovery of the stroke upper limbs still need to be explored. The main purpose of this research is to develop a smart phone with app system for stroke upper limb motor training, and further analyze its feasibility and treatment effects. The investigators randomly assigned chronic home stroke cases to the experimental group (n=20) and control group (n=20), each group received 8 weeks of treatment.

DETAILED DESCRIPTION:
Stroke rehabilitation (including occupational therapy and physical therapy) for stroke patients can enhance the upper and lower limb function, daily of daily activity improvement, and be beneficial to the family members' quality of life. Literature studies have supported the use of tele-rehabilitation to be as effective as stroke home rehabilitation. Stroke tele-rehabilitation model can use smartphones and apps to practice the mobile health model. This technology with remote rehabilitation have the important characteristics, including ease of use, high-intensity, repetitive exercises, and providing feedback information, to facilitate the recovery of training functions. Nevertheless, effects of tele-rehabilitation analysis for the proximal recovery of the stroke upper limbs still need to be explored. The main purpose of this research is to develop a smart phone with app system for stroke upper limb motor training, and further analyze its feasibility and treatment effects. The investigators randomly assigned chronic home stroke cases to the experimental group (n=20) and control group (n=20), each group received 8 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* First onset
* Unilateral Hemiplegia
* No obvious cognitive impairment (Mini-Mental State Examination (MMSE) score > 23)
* The FMA upper limb movement score is above 30 points
* Those who have used a smartphone for more than 3 months before the onset of the disease or at present
* Those who have no obvious vision loss and can read the text on mobile phones clearly
* Those who own a smart phone

Exclusion Criteria:

* Language barriers or aphasia
* Other orthopedic diseases (such as severe shoulder pain, joint contractures) or nerve damage (such as peripheral nerve damage) that affect the movement of the upper limbs
* Feel severe Absence, FMA sensory score <12 points
* Other progressive diseases such as cancer, amyotrophic lateral sclerosis, multiple sclerosis, etc

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-12-31 (Actual); Primary Completion 2020-06-18 (Actual); Study Completion 2021-03-26 (Actual)

PRIMARY OUTCOMES:
FUGL-MEYER ASSESSMENT-UE, FMA) | pre-test, post-test(Change from pre-test FUGL-MEYER ASSESSMENT-UE after 8 weeks' intervention)
  Fugl-Meyer Assessment (FMA) scale is an index to assess the sensorimotor impairment in individuals who have had stroke.
Box and Block Test | pre-test, post-test(Change from pre-test Box and Block Test after 8 weeks' intervention)
  The Box and Block Test (BBT) measures unilateral gross manual dexterity. It is a quick, simple and inexpensive test. It can be used with a wide range of populations, including clients with stroke.
Grip Strength Assessment | pre-test, post-test(Change from pre-test Grip Strength Assessment after 8 weeks' intervention)
  Grip strength is a measure of muscular strength or the maximum force/tension generated by one's forearm muscles. It can be used as a screening tool for the measurement of upper body strength and overall strength.
System Usability Scale | only post-test(after 8 weeks' intervention)
  The System Usability Scale, or SUS, is a simple survey that provides a high-level score for the usability of a product.
The Ruff 2 & 7 Selective Attention Test | pre-test, post-test(Change from pre-test The Ruff 2 & 7 Selective Attention Test after 8 weeks' intervention)
  The Ruff 2 and 7 Selective Attention Test (RSAT) is designed to measure selective attention.

CONTACTS AND LOCATIONS:
Overall Officials: Jyh-Jong Chang, PhD, Principal Investigator — Kaohsiung Medical University
Locations (1):
- Department of Occupational Therapy, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: starting one year after publication
Access Criteria: For Meta-analysis study

REFERENCES:
- [Result] Wu N, Gong E, Wang B, Gu W, Ding N, Zhang Z, Chen M, Yan LL, Oldenburg B, Xu LQ. A Smart and Multifaceted Mobile Health System for Delivering Evidence-Based Secondary Prevention of Stroke in Rural China: Design, Development, and Feasibility Study. JMIR Mhealth Uhealth. 2019 Jul 19;7(7):e13503. doi: 10.2196/13503. PMID 31325288
- See also: A Smart and Multifaceted Mobile Health System for Delivering Evidence-Based Secondary Prevention of Stroke in Rural China: Design, Development, and Feasibility Study — https://pubmed.ncbi.nlm.nih.gov/31325288/